CLINICAL TRIAL: NCT00003896
Title: Phase II Evaluation of Intravenous Paclitaxel, Intraperitoneal Cisplatin, Intravenous Liposomal Doxorubicin and Intraperitoneal Paclitaxel in Women With Optimally-Debulked Stage III Epithelial Ovarian Cancer
Brief Title: S9912 Combination Chemo in Stage III Ovarian Cancer,
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067066; S9912 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Cisplatin; liposomal doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel/cisplatin/Liposomal Doxorubicin (Experimental): paclitaxel, cisplatin and liposomal doxorubicin
  Interventions: Drug: cisplatin; Drug: liposomal doxorubicin; Drug: paclitaxel

INTERVENTIONS:
Drug: cisplatin
  Other Names: platinol
Drug: liposomal doxorubicin
  Other Names: pegylated liposomal doxorubicin hydrochloride; doxil
Drug: paclitaxel
  Other Names: taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel, cisplatin, and liposomal doxorubicin in treating women who have undergone surgery for stage III ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of intraperitoneal (IP) cisplatin, IP and IV paclitaxel, and IV doxorubicin HCl liposome, in terms of progression-free survival and overall survival, in patients with optimally debulked stage III ovarian epithelial, fallopian tube, or primary peritoneal cancer.
* Determine the feasibility of and toxic effects associated with this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours on day 1, intraperitoneal (IP) cisplatin over 30-60 minutes on day 2, IP paclitaxel over 30-60 minutes on day 8, and doxorubicin HCl liposome IV over 1 hour on day 8. Patients not able to tolerate IP infusion receive paclitaxel IV and cisplatin IV on day 1 only. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III ovarian epithelial, fallopian tube, or primary peritoneal carcinoma

  * Tumor involves one or both ovaries with microscopically confirmed peritoneal metastasis outside the pelvis and/or regional lymph node metastasis
  * No tumors of borderline or low malignant potential only
  * Mixed Mullerian tumors allowed
* Must have optimal disease defined as no residual lesions after resection or residual disease such that no single lesion measures greater than 1 cm in diameter
* Must have undergone staging exploratory laparotomy with tumor debulking within the past 70 days

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* SWOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 2 times ULN

Renal:

* Creatinine clearance ≥ 50 mL/min

Cardiovascular:

* No congestive heart failure
* No cardiac arrhythmia
* No myocardial infarction or unstable angina within the past 6 months
* Patients with a history of myocardial disease must not have ischemia or pathologic arrhythmias and must have an ejection fraction > 50% by MUGA

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active or uncontrolled infection
* No concurrent fever
* No grade 2 or greater sensory neuropathy
* No severe gastrointestinal symptoms (i.e., partial obstruction) and/or bleeding, diarrhea, or abdominal tenderness suggestive of peritoneal irritation or infection
* No erythema or tenderness of abdominal incision or port site suggestive of underlying infection
* No other malignancy within the past five years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for ovarian cancer

Chemotherapy:

* No prior chemotherapy for ovarian cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior pelvic radiotherapy for ovarian cancer

Surgery:

* See Disease Characteristics
* Recovered from all reversible surgery-related toxic effects

Other:

* No other concurrent antitumor treatment
* No concurrent antibiotics for infection of undetermined etiology

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 1999-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet O. Smith, MD, Study Chair — University of New Mexico Cancer Center
Locations (104):
- United States (104):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - University of California Davis Cancer Center, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Saint Rose Hospital, Hayward, California
  - Valley Memorial Hospital, Livermore, California
  - Highland General Hospital, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Cancer Care Center at Battle Creek Health System, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, East Lansing, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Mercy Hospital, Port Huron, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Judy L. Schmidt, MD, FACP, P. C., Missoula, Montana
  - Good Samaritan Health Systems, Kearney, Nebraska
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Harrington Cancer Center, Amarillo, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cancer Care Center at Skagit Valley Hospital, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Smith HO, Moon J, Wilczynski SP, Tiersten AD, Hannigan EV, Robinson WR, Rivkin SE, Anderson GL, Liu PY, Markman M. Southwest Oncology Group Trial S9912: intraperitoneal cisplatin and paclitaxel plus intravenous paclitaxel and pegylated liposomal doxorubicin as primary chemotherapy of small-volume residual stage III ovarian cancer. Gynecol Oncol. 2009 Aug;114(2):206-9. doi: 10.1016/j.ygyno.2009.04.023. Epub 2009 May 23. PMID 19464730

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel/CDDP/Lipo Doxorubicin: intravenous paclitaxel (day 1), intraperitoneal cisplatin (day 2), intraperitoneal paclitaxel and intravenous liposomal doxorubicin (day 8)
Period: Overall Study
Arm/Group | Paclitaxel/CDDP/Lipo Doxorubicin
Started | 68
Eligible | 63 (2 eligible patients did not have any toxicity assessments reported.)
Completed | 39
Not Completed | 29
Not completed — Adverse Event | 16
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Death | 3
Not completed — not protocol specified | 3
Not completed — ineligible | 5

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel/CDDP/Lipo Doxorubicin
Number analyzed (Participants) | 63
Age Continuous [Median (Full Range); unit: years] | 59 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 59
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: From date of registration to date of progression (as defined per RECIST), symptomatic deterioration or death due to any cause.
Time Frame: Once a month for 6 months, then every 6 months for up to 2 years, then annually thereafter.
Population: Eligible patients who began the treatment intervention
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/CDDP/Lipo Doxorubicin
Number analyzed (Participants) | 63
months | 25 [19 to 34]

2. Primary Outcome: Overall Survival
Description: from date of registration to date of death due to any cause. Patients last known to be alive wer censored at date of last contact
Time Frame: Weekly for 6 weeks, then every 6 months for 2 years, then annually thereafter.
Population: All eligible patients who began the treatment intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel/CDDP/Lipo Doxorubicin
Number analyzed (Participants) | 63
months | 51 [42 to 59]

3. Secondary Outcome: Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Weekly during 6 weeks of protocol treatment
Population: Paclitaxel/CDDP/Liposomal doxorubicin
Measure: Number; unit: Participants
Arm/Group | Paclitaxel/CDDP/Liposomal Doxorubicin
Number analyzed (Participants) | 61
Participants
  Abdominal pain/cramping | 7
  Allergic reaction | 2
  Anemia | 5
  Anorexia | 5
  Ataxia (incoordination) | 1
  Bone pain | 1
  Cardiac ischemia/infarction | 1
  Catheter related infection | 4
  Chest pain,not cardio or pleur | 1
  Confusion | 1
  Constipation/bowel obstruction | 5
  Creatinine increase | 1
  Dehydration | 5
  Diarrhea without colostomy | 4
  Dizziness/light headedness | 1
  Dyspepsia/heartburn | 1
  Dyspnea | 2
  Esophagitis/dysphagia | 1
  Fatigue/malaise/lethargy | 10
  Febrile neutropenia | 6
  GI Mucositis, NOS | 1
  GU fistula | 1
  Hand-foot skin reaction | 3
  Headache | 1
  Hyperglycemia | 2
  Hypertension | 1
  Hypoalbuminemia | 1
  Hypocalcemia | 1
  Hypokalemia | 4
  Hypomagnesemia | 2
  Hypotension | 1
  Ileus | 2
  Infection w/o 3-4 neutropenia | 5
  Infection with 3-4 neutropenia | 4
  Infection, unk ANC | 2
  Insomnia | 1
  Intestinal fistula | 1
  Leukopenia | 32
  Lymphopenia | 16
  Metabolic-other | 1
  Myalgia | 1
  Nausea | 14
  Neutropenia/granulocytopenia | 35
  PRBC transfusion | 5
  Platelet transfusion | 1
  Pneumonitis/infiltrates | 1
  Renal failure | 1
  Respiratory infect w/ neutrop | 2
  SGOT (AST) increase | 1
  SGPT (ALT) increase | 1
  Somnolence/consciousness loss | 1
  Stomatitis/pharyngitis | 4
  Thrombocytopenia | 5
  Thrombosis/embolism | 4
  Urinary tr infect w/o neutrop | 2
  Vomiting | 9
  Weakness (motor neuropathy) | 3
  Weight loss | 1

ADVERSE EVENTS:
Time Frame: Weekly until the end of 6 weeks of protocol treatment.
Arm/Group | Paclitaxel/CDDP/Liposomal Doxorubicin
Serious Adverse Events (participants affected / at risk) | 2/61
Other Adverse Events (participants affected / at risk) | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/CDDP/Liposomal Doxorubicin (N=61)
GI Mucositis, NOS (Gastrointestinal disorders) | 1
Infection with 3-4 neutropenia (Infections and infestations) | 1
Infection, unk ANC (Infections and infestations) | 1
Leukopenia (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/CDDP/Liposomal Doxorubicin (N=61)
Anemia (Blood and lymphatic system disorders) | 43
Febrile neutropenia (Blood and lymphatic system disorders) | 6
PRBC transfusion (Blood and lymphatic system disorders) | 5
Sinus tachycardia (Cardiac disorders) | 4
Inner ear-hearing loss (Ear and labyrinth disorders) | 4
Abdominal pain/cramping (Gastrointestinal disorders) | 38
Constipation/bowel obstruction (Gastrointestinal disorders) | 25
Diarrhea without colostomy (Gastrointestinal disorders) | 20
Dyspepsia/heartburn (Gastrointestinal disorders) | 5
Esophagitis/dysphagia (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 45
Stomatitis/pharyngitis (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 32
Edema (General disorders) | 4
Fatigue/malaise/lethargy (General disorders) | 38
Fever without neutropenia (General disorders) | 5
Pain-other (General disorders) | 7
Allergic reaction (Immune system disorders) | 5
Infection w/o 3-4 neutropenia (Infections and infestations) | 7
Catheter related infection (Injury, poisoning and procedural complications) | 7
Local injection site reaction (Injury, poisoning and procedural complications) | 6
Leukopenia (Investigations) | 51
Lymphopenia (Investigations) | 32
Neutropenia/granulocytopenia (Investigations) | 48
SGOT (AST) increase (Investigations) | 5
Thrombocytopenia (Investigations) | 21
Weight loss (Investigations) | 24
Anorexia (Metabolism and nutrition disorders) | 25
Dehydration (Metabolism and nutrition disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Dizziness/light headedness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 8
Sensory neuropathy (Nervous system disorders) | 23
Taste disturbance (Nervous system disorders) | 11
Weakness (motor neuropathy) (Nervous system disorders) | 6
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 39
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 14
Rash/desquamation (Skin and subcutaneous tissue disorders) | 17
Flushing (Vascular disorders) | 4
Hypotension (Vascular disorders) | 6
Thrombosis/embolism (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No